CLINICAL TRIAL: NCT02133196
Title: A Phase II Study Using Autologous Young Tumor-Infiltrating Lymphocytes Derived From Patients With Non-Small Cell Lung Cancer Following Non-Myeloablative Lymphocyte Depleting Preparative Regimen
Brief Title: T Cell Receptor Immunotherapy for Patients With Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140104; 14-C-0104
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2025-11-03

CONDITIONS: Advanced Non-Small Cell Lung Cancer; Squamous Cell Carcinoma; Advanced NSCLC; Adenosquamous Carcinoma; Adenocarcinoma
Keywords: Metastatic; Non-Small Cell Lung Cancer; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Adenosquamous; Adenocarcinoma; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — aldesleukin; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/High-Dose Aldesleukin (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine plus young TIL plus high-dose Aldesleukin
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL
- 2/Low-Dose Aldesleukin (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine plus young TIL plus low-dose Aldesleukin
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL

INTERVENTIONS:
Drug: Aldesleukin — Aldesleukin 720,000 (Arm 1) or 72,000 (Arm 2) IU/kg IV (based on total body weight) over 15 minutes every 8 hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to a maximum of 9 doses in Arm 1 and 12 doses in Arm 2.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with Mesna 15 mg/kg/day X 2 days over 1 hour.
Biological: Young TIL — Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.

SUMMARY:
Background:

The NCI Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 100 patients. In this study, we are selecting a specific subset of white blood cells from the tumor that we think are the most effective in fighting tumors and will use only these cells in making the tumor fighting cells.

Objective:

The purpose of this study is to see if these specifically selected tumor fighting cells can cause non-small cell lung cancer (NSCLC) tumors to shrink and to see if this treatment is safe.

Eligibility:

- Adults age 18-72 with NSCLC who have a tumor that can be safely removed.

Design:

* Work up stage: Patients will be seen as an outpatient at the NIH clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Surgery: If the patients meet all of the requirements for the study they will undergo surgery to remove a tumor that can be used to grow the TIL product.
* Leukapheresis: Patients may undergo leukapheresis to obtain additional white blood cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the TIL cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
Background:

* Patients with metastatic non-small cell lung cancer (NSCLC) have few approved therapeutic options and those that exist are of transient benefit.
* Recent clinical experiences with experimental agents that release checkpoints on the host immune response (such as anti-PD-1 and anti-PDL1 antibody) have induced tumor regressions in patients with NSCLC.
* Data from sequencing the genomes of human cancers have shown that, like malignant melanoma, NSCLC has a very high rate of tumor-specific genomic mutation.
* In metastatic melanoma, a tumor infiltrating lymphocyte cell therapy product (TIL) can mediate the regression of bulky disease at any site when administered to an autologous patient with high dose aldesleukin following a non-myeloablative but lymphodepleting chemotherapy preparative regimen.
* Recent studies on tumor infiltrating lymphocytes from melanoma have demonstrated that they can frequently recognize tumor-specific mutated proteins as "foreign" antigens and that is one hypothesis as to why melanoma is such an immunogenic tumor.
* We propose to investigate the feasibility, safety, and efficacy of growing and administering an autologous tumor infiltrating lymphocyte product (TIL) to patients with metastatic NSCLC

Objectives:

Primary objective:

-To determine the rate of tumor regression in patients with advanced non-small cell lung cancer (NSCLC) who receive an autologous tumor infiltrating lymphocyte product (TIL) plus aldesleukin following a lymphodepleting preparative regimen.

Eligibility:

* Patients who are >= 18 years of age and <= 72 years of age must have:

  * Advanced NSCLC refractory to standard therapy
  * A site of tumor that can be excised with minimal morbidity and mortality or that requires excision for clinical indications
  * At least one remaining site of measurable disease
  * Normal basic laboratory values.
* Patients may not have:

  * Concurrent major medical illnesses that preclude aldesleukin administration or immunosuppression;
  * Severe hepatic function impairment due to liver metastatic burden;
  * Any form of immunodeficiency;
  * Severe hypersensitivity to any of the agents used in this study;
  * Symptomatic brain metastases or more than 3 CNS metastases

Design:

* Patients will undergo biopsy or resection to obtain tumor for generation of autologous tumor infiltrating lymphocyte cultures and autologous cancer cell lines.
* The TIL product will be generated according to current TIL-lab standard operating procedures, using interleukin-2 and OKT3 antibody.
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine
* Cohort 1 will receive TIL on day 0 and then begin high-dose aldesleukin (720,000 IU/kg IV); cohort 2 will receive TIL on day 0 and then begin low-dose aldesleukin (72,000 IU/kg IV). Assignment to this cohort will be made if there are concomitant medical conditions that would preclude the use of high-dose aldesleukin
* Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion.
* For both cohorts 1 and 2, using a Phase II design, 21 patients will be initially enrolled in each group to assess toxicity and tumor responses. If two or more of the first 21 patients per group show a clinical response (PR or CR), accrual will continue to 41 patients, targeting a 20% goal for objective response. In order to allow for a small number of non evaluable patients, a total of 85 patients may be enrolled over 5 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic (stage IV) or unresectable non-small cell lung cancer (including but not limited to squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinomas) with at least one lesion that is resectable for TIL generation. (Note: neuroendocrine tumors are not eligible.)
  2. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
  3. All patients must have had at least one appropriate first line systemic therapy and progressed.
  4. Clinical performance status of ECOG 0 or 1.
  5. Age >= 18 years of age and <= 72 years of age.
  6. Patients of both sexes must be willing to practice birth control from the time of enrollment on this study and for 12 months after the last dose of combined chemotherapy for individuals of childbearing potential (IOCBP) and for four months after treatment for individuals able to father a child.
  7. Willing to sign a durable power of attorney
  8. Able to understand and sign the Informed Consent Document

I. Hematology:

* Absolute neutrophil count > 1000/mm^3 without support of filgrastim
* Normal WBC (>= 2500/mm^3).
* Hemoglobin > 8.0 g/dl. Subjects may be transfused to reach this cut-off.
* Platelet count >= 80,000/mm^3

  j. Serology:
* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

  k. Chemistry:
* Serum ALT/AST <= 2.5 times the upper limit of normal.
* Serum creatinine <= 1.6 mg/dl.
* Total bilirubin <= 2 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin <= 3 mg/dl.

  l. IOCBP must have a negative pregnancy test or evidence that they are not pregnant (e.g., ultrasound or serial HCG measurements) prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.

  m. Patients must have completed any prior systemic therapy at the time of enrollment.

Note: Patients may have undergone minor surgical procedures or local radiotherapy within the past 4 weeks, as long as related major organ toxicities have recovered to grade 1 or less.

n. More than two weeks must have elapsed since any prior palliation for major bronchial occlusion or bleeding at the time the patient receives the preparative regimen, and patient's toxicities must have recovered to a grade 1 or less.

o. Subjects must be co-enrolled in protocol 03-C-0277.

EXCLUSION CRITERIA:

1. Participants who are nursing because of the potentially dangerous effects of the treatment on the infant.
2. Ongoing need for pharmacological immunosuppression, including steroids
3. Active systemic infections (e.g.: requiring anti-infective treatment), coagulation disorders or any other active or uncompensated major medical illnesses
4. Major bronchial occlusion or bleeding not amenable to palliation.
5. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency

   Disease and AIDS).
6. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. For select patients with a clinical history prompting cardiac evaluation: last known LVEF <= 45%.
9. For select patients with a clinical history prompting pulmonary evaluation: known FEV1 <= 50%
10. Any of the following will exclude patients from the high-dose aldesleukin arm, but may be eligible for the low-dose aldesleukin arm:

    * Greater than 2 invasive thoracic procedures
    * Poor exercise tolerance
    * Greater than 66 years of age
    * Clinically significant patient history which in the judgment of the Principal Investigator would compromise the patient s ability to tolerate high-dose.
11. Patients who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2014-10-23 (Actual); Primary Completion 2027-10-23 (Estimated); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who have a clinical response to treatment (objective tumor regression)

SECONDARY OUTCOMES:
Phenotypic and functional characteristics of TIL | 2-4 years post cell infusion
  Find in vitro characteristics of the infused cells which correlate with in vivo antitumor activity. Evaluation of the activity, specificity, and telomere length of infused TIL.
Frequency and severity of treatment-related adverse events | 30 days after end of treatment
  Aggregate of all adverse events, as well as their frequency and severity
Feasibility of generating TIL from patients with NSCLC | 3-6 months post cell harvest

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Delbaldo C, Michiels S, Rolland E, Syz N, Soria JC, Le Chevalier T, Pignon JP. Second or third additional chemotherapy drug for non-small cell lung cancer in patients with advanced disease. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD004569. doi: 10.1002/14651858.CD004569.pub2. PMID 17943820
- [Background] Boni C, Tiseo M, Boni L, Baldini E, Recchia F, Barone C, Grossi F, Germano D, Matano E, Marini G, Labianca R, Di Costanzo F, Bagnulo A, Pennucci C, Caroti C, Mencoboni M, Zanelli F, Prochilo T, Cafferata MA, Ardizzoni A; Gruppo Oncologico Italiano di Ricerca Clinica (GOIRC). Triplets versus doublets, with or without cisplatin, in the first-line treatment of stage IIIB-IV non-small cell lung cancer (NSCLC) patients: a multicenter randomised factorial trial (FAST). Br J Cancer. 2012 Feb 14;106(4):658-65. doi: 10.1038/bjc.2011.606. Epub 2012 Jan 12. PMID 22240782
- [Derived] Malekzadeh P, Pasetto A, Robbins PF, Parkhurst MR, Paria BC, Jia L, Gartner JJ, Hill V, Yu Z, Restifo NP, Sachs A, Tran E, Lo W, Somerville RP, Rosenberg SA, Deniger DC. Neoantigen screening identifies broad TP53 mutant immunogenicity in patients with epithelial cancers. J Clin Invest. 2019 Mar 1;129(3):1109-1114. doi: 10.1172/JCI123791. Epub 2019 Feb 4. No abstract available. PMID 30714987
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-C-0104.html